CLINICAL TRIAL: NCT05989516
Title: Cyst Extraction With Pericyst Reduction and Omentopexy as a Treatment of Choice for Hydatid Liver Disease Caused by E. Granulosus: Retrospective Observational Review of a Single Center Experience
Brief Title: Surgical Treatment of Hydatid Liver Disease
Status: Completed | Type: Observational
Sponsor: University Hospital for Surgical Diseases St. Naum Ohridsk i- Skopje (Other)
Responsible Party: Principal Investigator, Elena Zafirovikj, Dr., University Hospital for Surgical Diseases St. Naum Ohridsk i- Skopje
Other Study IDs: 001/0/2023
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Hydatid Cyst, Hepatic
MeSH Terms: conditions — Echinococcosis, Hepatic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to show that cyst extraction with pericyst reduction and omentopexy is a suitable treatment for liver hydatid disease caused by E.Granulossus with a low rate of complication and recurrence.

ELIGIBILITY:
Inclusion Criteria:

* hydatid liver disease

Exclusion Criteria:

* hydatid disease present outside the liver

Ages: 16 Years to 99 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: We have analyzed 72 patients diagnosed with liver hydatid disease for a period of 10 years from January 2006 until January 2017 treated surgically by cyst extraction, pericystectomy, and omentopexy.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Post operative complications | one month
  Listing of complications according to Clavien -Dindo classification

SECONDARY OUTCOMES:
Recurrence rate | 5 years
  Recurrence rate of hydatid disease in patients

CONTACTS AND LOCATIONS:
Overall Officials: Elena Zafirovikj, MD, Principal Investigator — UHSD St. Naum Ohridski
Locations (1):
- Elena Zafirovikj, Skopje, North Macedonia

IPD SHARING:
Plan to Share IPD: Undecided